CLINICAL TRIAL: NCT01774968
Title: Two Treatment Approaches for Human Regular U-500 Insulin (Thrice-Daily Versus Twice-Daily) in Subjects With Type 2 Diabetes Mellitus Not Achieving Adequate Glycemic Control on High-Dose U-100 Insulin Therapy With or Without Oral Agents: A Randomized, Open-Label, Parallel Clinical Trial
Brief Title: Study of Human Regular U-500 Insulin in Adult Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14838; B5K-US-IBHC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Regular U-500 Insulin TID (Experimental): Human Regular U-500 Insulin (U-500R) titrated based on blood glucose readings, administered subcutaneously (SC), three times a day (TID) for 24 weeks.
  Interventions: Drug: Human Regular U-500 Insulin
- Human Regular U-500 Insulin BID (Experimental): U-500R Insulin titrated based on blood glucose readings, administered SC, two times a day (BID) for 24 weeks.
  Interventions: Drug: Human Regular U-500 Insulin

INTERVENTIONS:
Drug: Human Regular U-500 Insulin
  Other Names: LY041001; Humulin R; U-500R

SUMMARY:
The main purpose of this study is to compare the effectiveness of Human Regular U-500 Insulin three times a day versus twice a day.

ELIGIBILITY:
Major Inclusion Criteria:

* Have type 2 diabetes mellitus (World Health Organization [WHO] Classification of Diabetes)
* Have a body mass index (BMI) ≥25 kilogram per square meter (kg/m^2)
* Have Glycated Hemoglobin A1c (HbA1c) ≥7.5% and ≤12.0%, as measured by the central laboratory at entry
* Current U-100 insulin/analogue users on >200 and ≤600 units per day for ≥3 months at study entry and reconfirmed at randomization
* Have a history of stable body weight for at least 3 months prior to study entry
* Concomitant medications may include metformin (MET), dipeptidyl peptidase-4 (DPP-4) inhibitors approved for use with insulin at time of study entry (for example, sitagliptin, saxagliptin, and linagliptin), pioglitazone, and/or sulfonylureas (SUs)/glinides (repaglinide or nateglinide). Participant's oral antihyperglycemic drug (OAD) dose(s) must have been stable for ≥3 months

Major Exclusion Criteria:

* Have type 1 diabetes mellitus or other types of diabetes mellitus apart from type 2 diabetes mellitus
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine aminotransferase or aspartate aminotransferase levels ≥3 times the upper limit of the reference range
* Have chronic kidney disease stage 4 and higher or history of renal transplantation
* Have history of more than 1 episode of severe hypoglycemia within the 6 months prior to study entry
* Have received insulin by continuous subcutaneous insulin infusion in the 3 months prior to study entry
* Have received U-500R in the 3 months prior to study entry
* Have had a blood transfusion or severe blood loss within 3 months prior to study entry or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia
* Are taking chronic systemic glucocorticoid therapy or have received such therapy within the 4 weeks immediately prior to study entry
* Have an irregular sleep/wake cycle
* Have used rosiglitazone, once- or twice-daily glucagon-like peptide-1 (GLP-1) receptor agents, pramlintide, or other injectable or oral antihyperglycemic therapy not listed in the inclusion criteria in the 3 months prior to study entry. Participants may not have used once-weekly GLP-1 receptor agents in the 4 months prior to study entry
* Have used any weight loss drugs in the 3 months prior to study entry
* Have a history of bariatric surgery
* Have a history of malignancy other than basal cell or squamous cell skin cancer
* Have New York Heart Association (NYHA) Class III or IV per NYHA Cardiac Disease Functional Classification
* Are breastfeeding or pregnant, or intend to become pregnant during the course of the study, or are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (39):
- United States (35):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crystal Lake, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaumont, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Lomas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- [Derived] Kabul S, Hood RC, Duan R, DeLozier AM, Settles J. Patient-reported outcomes in transition from high-dose U-100 insulin to human regular U-500 insulin in severely insulin-resistant patients with type 2 diabetes: analysis of a randomized clinical trial. Health Qual Life Outcomes. 2016 Sep 30;14(1):139. doi: 10.1186/s12955-016-0541-4. PMID 27716283
- [Derived] Mari A, Rosenstock J, Ma X, Li YG, Jackson JA. OPTIMIZED HUMAN REGULAR U-500 INSULIN TREATMENT IMPROVES beta-CELL FUNCTION IN SEVERELY INSULIN-RESISTANT PATIENTS WITH LONG-STANDING TYPE 2 DIABETES AND HIGH INSULIN REQUIREMENTS. Endocr Pract. 2015 Dec;21(12):1344-52. doi: 10.4158/EP15898.OR. Epub 2015 Aug 26. PMID 26307903
- [Derived] Hood RC, Arakaki RF, Wysham C, Li YG, Settles JA, Jackson JA. TWO TREATMENT APPROACHES FOR HUMAN REGULAR U-500 INSULIN IN PATIENTS WITH TYPE 2 DIABETES NOT ACHIEVING ADEQUATE GLYCEMIC CONTROL ON HIGH-DOSE U-100 INSULIN THERAPY WITH OR WITHOUT ORAL AGENTS: A RANDOMIZED, TITRATION-TO-TARGET CLINICAL TRIAL. Endocr Pract. 2015 Jul;21(7):782-93. doi: 10.4158/EP15612.OR. Epub 2015 Mar 26. PMID 25813411

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Started | 162 | 163
Received at Least 1 Dose of Study Drug | 162 | 161
Completed | 132 | 128
Not Completed | 30 | 35
Not completed — Adverse Event | 4 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 5 | 1
Not completed — Protocol Violation | 14 | 13
Not completed — Sponsor Decision | 0 | 2
Not completed — Withdrawal by Subject | 6 | 11

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Human Regular U-500 Insulin TID: U-500R Insulin titrated based on blood glucose readings, administered SC, TID for 24 weeks.
- Human Regular U-500 Insulin BID: U-500R Insulin titrated based on blood glucose readings, administered SC, BID for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID | Total
Number analyzed (Participants) | 162 | 163 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.31 (10.51) | 55.50 (9.03) | 55.41 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 74 | 153
  Male | 83 | 89 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 30 | 62
  Not Hispanic or Latino | 130 | 133 | 263
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 21 | 19 | 40
  White | 133 | 133 | 266
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 146 | 149 | 295
  Puerto Rico | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Glycated Hemoglobin A1c (HbA1c)
Description: Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with investigator, baseline total daily dose (TDD; ≤300 or >300 units), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline HbA1c as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
percentage of HbA1c | -1.12 (0.08) | -1.22 (0.08)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin TID vs Human Regular U-500 Insulin BID; Approximately 325 participants were to be randomized (in a 1:1 ratio of U-500R insulin TID:BID) and 260 were to complete the study (with a 20% dropout rate). The 260 completers would provide a 66.4% chance to show equivalence of TID and BID algorithms, 14.4% chance to show noninferiority of TID, 2.5% chance to superiority of TID, 14.4% chance to show noninferiority of BID, and 2.5% chance to show superiority of BID, assuming a difference in HbA1c change of 0% and a standard deviation of 1.1%; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p = 0.3709, Mixed Models Analysis; LS Mean Difference = -0.10, 95% CI 2-sided [-0.33 to 0.12]

2. Secondary Outcome: Percentage of Participants Achieving HbA1c of ≤6.5%, <7.0%, <7.5%, and <8.0% at Week 24
Description: The percentage of participants achieving an HbA1c of ≤6.5%, <7.0%, <7.5%, and <8.0% at Week 24 was calculated by the dividing the number of participants meeting the criteria by the total number of participants analyzed, multiplied by 100.
Time Frame: Week 24
Population: Randomized participants who received at least 1 dose of U-500R, who were not at the HbA1c target at baseline, and had evaluable HbA1c data.
Measure: Number; unit: percentage of participants
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 159 | 161
percentage of participants
  HbA1c ≤6.5% (n=159, 161) | 20.13 | 23.60
  HbA1c <7.0% (n=158, 159) | 42.41 | 41.51
  HbA1c <7.5% (n=148, 143) | 64.19 | 61.54
  HbA1c <8.0% (n=120, 123) | 77.50 | 77.24

3. Secondary Outcome: 30-Day Adjusted Rate of Hypoglycemic Events
Description: Hypoglycemic events (HE) were classified as severe (an event requiring assistance from another person [accompanied by neurologic/cognitive impairment]), documented symptomatic (an event which is associated with signs/symptoms of hypoglycemia and plasma glucose [PG] ≤70 milligrams per deciliter [mg/dL]), documented symptomatic nocturnal (any documented symptomatic HE that occurred between bedtime and waking), or asymptomatic (any measured PG ≤70 mg/dL not accompanied by hypoglycemic signs/symptoms). The 30-day adjusted rate of HE is summarized cumulatively at 24 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Week 24
Population: Randomized participants who received at least 1 dose of U-500R.
Measure: Mean (Standard Deviation); unit: events per participant per 30 days
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
events per participant per 30 days
  Severe HE | 0.004 (0.028) | 0.009 (0.053)
  Documented Symptomatic HE | 3.343 (3.174) | 3.885 (3.448)
  Documented Symptomatic Nocturnal HE | 1.013 (1.438) | 1.299 (1.540)
  Asymptomatic HE | 1.340 (3.215) | 1.028 (2.231)

4. Secondary Outcome: Change From Baseline to Week 24 in Body Weight
Description: LS means of change from baseline were calculated using MMRM with investigator, baseline HbA1c (≤8% or >8%), baseline TDD (≤300 or >300 units), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline body weight as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
kilograms (kg) | 5.44 (0.41) | 4.88 (0.41)

5. Secondary Outcome: Change From Baseline to Week 24 in Total Daily Dose (TDD; Units) of Insulin
Description: Baseline TDD was defined as the last U-100 insulin TDD prior to receiving the first dose of U-500R insulin. LS means of change from baseline were calculated using MMRM with investigator, baseline HbA1c (≤8% or >8%), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline TDD as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable TDD data.
Measure: Least Squares Mean (Standard Error); unit: units
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
units | 55.19 (10.16) | 51.39 (10.24)

6. Secondary Outcome: Change From Baseline to Week 24 in Total Daily Dose (TDD; Units/kg) of Insulin
Description: as for outcome 5
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable TDD data.
Measure: Least Squares Mean (Standard Error); unit: units per kilogram (units/kg)
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
units per kilogram (units/kg) | 0.32 (0.08) | 0.32 (0.08)

7. Secondary Outcome: Change From Baseline to Week 24 in Fasting Plasma Glucose (FPG) Levels
Description: LS means of change from baseline were calculated using MMRM with investigator, baseline HbA1c (≤8% or >8%), baseline TDD (≤300 or >300 units), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline FPG as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable FPG data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 161 | 159
milligrams per deciliter (mg/dL) | -6.66 (5.64) | -8.86 (5.72)

8. Secondary Outcome: Time to Reach HbA1c Target Values
Description: The cumulative number of participants achieving an HbA1c of ≤6.5%, <7.0%, <7.5%, and <8.0% is summarized at Weeks 6, 12, 18, and 24. The number of participants at risk (n) is also provided for each target value and timepoint.
Time Frame: Baseline through 6, 12, 18, and 24 weeks.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 154 | 155
participants
  HbA1c ≤6.5%, Week 6 (n=154, 155) | 1 | 6
  HbA1c ≤6.5%, Week 12 (n=145, 151) | 15 | 15
  HbA1c ≤6.5%, Week 18 (n=140, 145) | 24 | 27
  HbA1c ≤6.5%, Week 24 (n=76, 65) | 28 | 37
  HbA1c <7.0%, Week 6 (n=154, 153) | 14 | 10
  HbA1c <7.0%, Week 12 (n=148, 149) | 31 | 36
  HbA1c <7.0%, Week 18 (n=144, 145) | 52 | 55
  HbA1c <7.0%, Week 24 (n=53, 52) | 60 | 65
  HbA1c <7.5%, Week 6 (n=144, 137) | 30 | 20
  HbA1c <7.5%, Week 12 (n=140, 134) | 59 | 59
  HbA1c <7.5%, Week 18 (n=136, 132) | 81 | 78
  HbA1c <7.5%, Week 24 (n=34, 31) | 90 | 87
  HbA1c <8.0%, Week 6 (n=117, 117) | 32 | 34
  HbA1c <8.0%, Week 12 (n=114, 115) | 66 | 72
  HbA1c <8.0%, Week 18 (n=111, 113) | 85 | 86
  HbA1c <8.0%, Week 24 (n=20, 19) | 89 | 95

9. Secondary Outcome: Percentage of Participants With Hypoglycemic Events
Description: Hypoglycemic events (HE) were classified as severe (an event requiring assistance from another person [accompanied by neurologic/cognitive impairment]), documented symptomatic (an event which is associated with signs/symptoms of hypoglycemia and plasma glucose [PG] ≤70 milligrams per deciliter [mg/dL]), documented symptomatic nocturnal (any documented symptomatic HE that occurred between bedtime and waking), or asymptomatic (any measured PG ≤70 mg/dL not accompanied by hypoglycemic signs/symptoms). The percentage of participants with HE at 24 weeks was calculated by the dividing the number of participants meeting the criteria by the total number of participants analyzed, multiplied by 100. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Week 24
Population: Randomized participants who received at least 1 dose of U-500R.
Measure: Number; unit: percentage of participants
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
percentage of participants
  Severe HE | 1.85 | 3.73
  Documented Symptomatic HE | 91.98 | 90.06
  Documented Symptomatic Nocturnal HE | 77.78 | 80.75
  Asymptomatic HE | 64.20 | 66.46

10. Secondary Outcome: Change From Baseline to Week 24 in Number of Insulin Injections
Description: The number of insulin injections per day at baseline (Week 0) and at Week 24 are presented.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R. Last observation carried forward (LOCF) was used to impute missing postbaseline values.
Measure: Mean (Standard Deviation); unit: injections per day
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
injections per day
  Baseline | 4.765 (1.234) | 4.783 (1.307)
  Week 24 | 3.000 (0.000) | 2.000 (0.000)

11. Secondary Outcome: Mean Change From Baseline to Week 24 in 7-Point Self-Monitored Blood Glucose (SMBG)
Description: The 7-point SMBG is a participant self-administered blood glucose test which utilizes measurements at specific time points over a 24-hour period, including pre-morning meal (fasting), 2 hours after morning meal, pre-midday meal, 2 hours after midday meal, pre-evening meal, 2 hours after evening meal, and 3 AM. LS means of change from baseline were calculated using MMRM with investigator, baseline HbA1c (≤8% or >8%), baseline TDD (≤300 or >300 units), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline SMBG as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable SMBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 150 | 149
mg/dL
  Pre-morning Meal (n=150, 149) | -24.10 (3.96) | -29.19 (3.91)
  2 Hours After Morning Meal (n=146, 133) | -21.68 (4.29) | -31.32 (4.29)
  Pre-midday Meal (n=150, 149) | -23.54 (4.17) | -32.26 (4.11)
  2 Hours After Midday Meal (n=143, 133) | -24.31 (4.50) | -22.53 (4.49)
  Pre-evening Meal (n=150, 149) | -34.17 (3.93) | -32.96 (3.85)
  2 Hours After Evening Meal (n=147, 142) | -40.56 (4.13) | -38.36 (4.11)
  3 AM (n=147, 140) | -36.77 (4.34) | -47.82 (4.29)

12. Secondary Outcome: Change From Baseline to Week 24 in HbA1c Based on Baseline TDD Insulin ≤2.0 Units/kg and >2.0 Units/kg
Description: Participants were stratified by their baseline TDD insulin (≤2.0 units/kg or >2.0 units/kg). LS means of change from baseline were calculated using MMRM with investigator, baseline TDD (≤300 or >300 units), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline HbA1c as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
percentage of HbA1c
  Baseline TDD ≤2.0 units/kg (n=50, 46) | -0.99 (0.14) | -1.32 (0.15)
  Baseline TDD >2.0 units/kg (n=112, 115) | -1.19 (0.10) | -1.18 (0.10)

13. Secondary Outcome: Change From Baseline to Week 24 in 30-Day Adjusted Rate of Hypoglycemic Events Based on Baseline TDD Insulin ≤2.0 Units/kg and >2.0 Units/kg
Description: Participants were stratified by their baseline TDD insulin (≤2.0 units/kg or >2.0 units/kg). Hypoglycemic events (HE) were classified as severe (an event requiring assistance from another person [accompanied by neurologic/cognitive impairment]), documented symptomatic (DS; an event which is associated with signs/symptoms of hypoglycemia and plasma glucose [PG] ≤70 milligrams per deciliter [mg/dL]), or nocturnal (Noc; any documented symptomatic HE that occurred between bedtime and waking). The 30-day adjusted rate of HE is summarized cumulatively at 24 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R.
Measure: Mean (Standard Deviation); unit: events per participant per 30 days
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
events per participant per 30 days
  Severe HE, TDD ≤2 units/kg, Baseline (n=50, 46) | 0 (0) | 0 (0)
  Severe HE, TDD ≤2 units/kg, Week 24 (n=50, 46) | 0.004 (0.025) | 0 (0)
  Severe HE, TDD >2 units/kg, Baseline (n=112, 115) | 0 (0) | 0 (0)
  Severe HE, TDD >2 units/kg, Week 24 (n=112, 115) | 0.004 (0.029) | 0.013 (0.062)
  DS HE, TDD ≤2 units/kg, Baseline (n=50, 46) | 1.958 (4.808) | 1.454 (3.251)
  DS HE, TDD ≤2 units/kg, Week 24 (n=50, 46)) | 2.356 (2.352) | 3.131 (3.204)
  DS HE, TDD >2 units/kg, Baseline (n=112, 115) | 2.037 (4.382) | 1.730 (3.180)
  DS HE, TDD >2 units/kg, Week 24 (n=112, 115) | 3.784 (3.397) | 4.186 (3.509)
  Noc. HE, TDD ≤2 units/kg, Baseline (n=50, 46) | 1.066 (2.045) | 0.711 (1.965)
  Noc. HE, TDD ≤2 units/kg, Week 24 (n=50, 46) | 1.105 (1.153) | 1.282 (1.431)
  Noc. HE, TDD >2 units/kg, Baseline (n=112, 115) | 0.792 (2.465) | 0.585 (1.445)
  Noc. HE, TDD >2 units/kg, Week 24 (n=112, 115) | 1.522 (2.018) | 1.753 (1.934)

14. Secondary Outcome: Change From Baseline to Week 24 in Percentage of Participants With Hypoglycemic Events Based on Baseline TDD Insulin ≥2.0 Units/kg and <2.0 Units/kg
Description: Participants were stratified by their baseline TDD insulin (≤2.0 units (U)/kg or >2.0 U/kg). The percentage of participants at risk of developing hypoglycemia (including documented symptomatic, asymptomatic, probable symptomatic, unspecified, or severe hypoglycemia) is presented at Baseline and at Week 24 and was calculated using MMRM fit with options of the binomial distribution and log link function including treatment, TDD (>300 units or ≤300 units), pioglitazone use (yes or no), visit, and treatment-by-visit interaction as fixed effects, and baseline HbA1c value as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R.
Measure: Number; unit: percentage of participants
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
percentage of participants
  Baseline TDD≤2.0 U/kg, Baseline risk (n=50, 46) | 56.00 | 39.13
  Baseline TDD ≤2.0 U/kg, Week 24 risk (n=50, 46) | 94.00 | 86.96
  Baseline TDD >2.0 U/kg, Baseline risk (n=112, 115) | 47.32 | 51.30
  Baseline TDD >2.0 U/kg, Week 24 risk (n=112, 115) | 96.43 | 97.39

15. Secondary Outcome: Change From Baseline to Week 24 in Body Weight Based on Baseline TDD Insulin ≥2.0 Units/kg and <2.0 Units/kg
Description: Participants were stratified by their baseline TDD insulin (≤2.0 units/kg or >2.0 units/kg). LS means of change from baseline were calculated using MMRM with investigator, baseline HbA1c (≤8% or >8%), baseline TDD (≤300 or >300 units), treatment (TID or BID), visit, and treatment-by-visit interaction as fixed effects and baseline body weight as a covariate.
Time Frame: Baseline, Week 24
Population: Randomized participants who received at least 1 dose of U-500R with evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Number analyzed (Participants) | 162 | 161
kg
  Baseline TDD insulin ≤2.0 units/kg (n=50, 46) | 6.11 (0.88) | 6.09 (0.93)
  Baseline TDD insulin >2.0 units/kg (n=112, 115) | 5.08 (0.44) | 4.40 (0.43)

ADVERSE EVENTS:
Description: The Serious Adverse Events and Other Adverse Events Tables include all randomized participants.
Arm/Group | Human Regular U-500 Insulin TID | Human Regular U-500 Insulin BID
Serious Adverse Events (participants affected / at risk) | 28/162 | 27/163
Other Adverse Events (participants affected / at risk) | 80/162 | 94/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Regular U-500 Insulin TID (N=162) | Human Regular U-500 Insulin BID (N=163)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (2)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 1 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 1 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Regular U-500 Insulin TID (N=162) | Human Regular U-500 Insulin BID (N=163)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 10 (10)
Nausea (Gastrointestinal disorders) | 4 (4) | 9 (9)
Vomiting (Gastrointestinal disorders) | 4 (4) | 11 (11)
Oedema peripheral (General disorders) | 6 (6) | 10 (10)
Bronchitis (Infections and infestations) | 9 (9) | 5 (5)
Nasopharyngitis (Infections and infestations) | 13 (13) | 17 (17)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (10)
Headache (Nervous system disorders) | 13 (13) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days